CLINICAL TRIAL: NCT01973608
Title: A Safety Study for MSB0010445 in Combination With Stereotactic Body Radiation in Advanced Melanoma Subjects Following Prior Treatment With Ipilimumab
Brief Title: MSB0010445 and Stereotactic Body Radiation Therapy in Advanced Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is terminated prematurely as the sponsor decided to discontinue program of NHS-IL2 [MSB0010445]
Sponsor: EMD Serono (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 062235-005
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Melanoma
Keywords: Melanoma; MSB0010445; Dose limiting toxicity; Stereotactic body radiation therapy
MeSH Terms: conditions — Melanoma | interventions — Radiosurgery

ARMS (4):
- MSB0010445 Low Dose Cohort 0.3 mg/kg (Experimental)
  Interventions: Drug: MSB0010445 (0.3 milligram per kilogram [mg/kg]); Radiation: Stereotactic Body Radiation Therapy (SBRT)
- MSB0010445 Intermediate Dose Cohort 1.0 mg/kg (Experimental)
  Interventions: Drug: MSB0010445 (1.0 mg/kg); Radiation: Stereotactic Body Radiation Therapy (SBRT)
- MSB0010445 High Dose Cohort 1.8 mg/kg (Experimental)
  Interventions: Drug: MSB0010445 (1.8 mg/kg); Radiation: Stereotactic Body Radiation Therapy (SBRT)
- MSB0010445 High Dose Cohort 2.4 mg/kg (Experimental)
  Interventions: Drug: MSB0010445 (2.4 mg/kg); Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: MSB0010445 (0.3 milligram per kilogram [mg/kg]) — MSB0010445 will be administered at a single dose of 0.3 mg/kg as intravenous (IV) infusion over approximately 1 hour every 3 weeks (q3w) for the first 12 Weeks as a part of induction phase followed by maintenance dose of 0.3 mg/kg drug every three weeks until significant clinical progression, occurrence of unacceptable toxicity, or withdrawal of consent. The first administration of MSB0010445 will be performed 3 days after the last dose of Stereotactic Body Radiation Therapy (SBRT) to the targeted reference lesion.
  Arms: MSB0010445 Low Dose Cohort 0.3 mg/kg
Drug: MSB0010445 (1.0 mg/kg) — MSB0010445 will be administered at a single dose of 1.0 mg/kg as IV infusion over approximately 1 hour q3w for the first 12 Weeks as a part of induction phase followed by maintenance dose of 0.3 mg/kg drug every three weeks until significant clinical progression, occurrence of unacceptable toxicity, or withdrawal of consent. The first administration of MSB0010445 will be performed 3 days after the last dose of SBRT to the targeted reference lesion.
  Arms: MSB0010445 Intermediate Dose Cohort 1.0 mg/kg
Drug: MSB0010445 (1.8 mg/kg) — MSB0010445 will be administered at a single dose of 1.8 mg/kg as IV infusion over approximately 1 hour q3w for the first 12 Weeks as a part of induction phase followed by maintenance dose of 0.3 mg/kg drug every three weeks until significant clinical progression, occurrence of unacceptable toxicity, or withdrawal of consent. The first administration of MSB0010445 will be performed 3 days after the last dose of SBRT to the targeted reference lesion.
  Arms: MSB0010445 High Dose Cohort 1.8 mg/kg
Drug: MSB0010445 (2.4 mg/kg) — MSB0010445 will be administered at a single dose of 2.4 mg/kg as IV infusion over approximately 1 hour q3w for the first 12 Weeks as a part of induction phase followed by maintenance dose of 0.3 mg/kg drug every three weeks until significant clinical progression, occurrence of unacceptable toxicity, or withdrawal of consent. The first administration of MSB0010445 will be performed 3 days after the last dose of SBRT to the targeted reference lesion.
  Arms: MSB0010445 High Dose Cohort 2.4 mg/kg
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT will be administered using a dose and schedule recommended based upon the data showing the best abscopal effect using multiple fractions if one site will be targeted subject received 3 fractions (1 per day) of 8 Gray (Gy) each (total: 24 Gy). If the target lesion will be located in the thorax, the maximum total dose administered will be 18 Gy (3 x 6 Gy).

SUMMARY:
This is a Phase 2a, open-label, parallel group, partly randomized dose escalation trial to assess the safety and efficacy of a low dose, an intermediate dose, and high dose MSB0010445 given by intravenous infusion to subjects with advanced (unresectable or metastatic) melanoma in combination with stereotactic body radiation therapy (SBRT).

ELIGIBILITY:
Inclusion Criteria:

* Advanced unresectable or metastatic melanoma, previously treated with ipilimumab; anti-melanoma treatments, including anti-PD/PD-L1 or any other immunotherapy, are allowed provided no treatment from last dose of that treatment to trial enrolment
* Subjects need to have

  * one lesion that can be irradiated
  * at least 1 measurable lesion outside the radiation field, different from the lesion that will be irradiated
  * one lesion that can be biopsied before treatment with SBRT and MSB0010445
  * one lesion outside the radiation field that can be biopsied while on treatment with MSB0010445
* The lesion that is biopsied at Baseline can be the lesion that will be irradiated
* The lesion that will be biopsied while on treatment should not be a lesion that has been irradiated or biopsied at Baseline
* Signed written informed consent
* Male and female subjects at least 18 years of age
* Life expectancy greater than or equal to (>=) 4 months
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Active central nervous system metastasis
* Treatment with systemic anti-cancer therapy within the 30 days before the first dose of SBRT
* Pre-existing pericardial effusion or history of Grade >=2 pleural effusion or ascites within 3 months before first dose of SBRT
* Concurrent systemic therapy with steroids or other immunosuppressive agents except short-term systemic steroids for allergic reactions
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, Inc., Rockland MA, a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (1):
- Please Contact U.S. Medical Information, Rockland, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/Last subject (informed consent): 24 January 2014/17 December 2014. Study completion date:10 June 2015. The study was conducted at 6 sites in the United States.
Groups:
- MSB0010445 Low Dose Cohort 0.3 mg/kg: MSB0010445 was administered at a single dose of 0.3 mg/kg as intravenous (IV) infusion over approximately 1 hour every 3 weeks (q3w) for the first 12 Weeks as a part of induction phase followed by maintenance dose of 0.3 mg/kg drug every three weeks until significant clinical progression, occurrence of unacceptable toxicity, or withdrawal of consent. The first administration of MSB0010445 was performed 3 days after the last dose of Stereotactic Body Radiation Therapy (SBRT) to the targeted reference lesion. SBRT was administered using a dose and schedule recommended based upon the data showing the best abscopal effect using multiple fractions if one site was targeted subject received 3 fractions (1 per day) of 8 Gray (Gy) each (total: 24 Gy). If the target lesion was located in the thorax, the maximum total dose administered was 18 Gy (3 x 6 Gy).
- MSB0010445 Intermediate Dose Cohort 1.0 mg/kg: MSB0010445 was administered at a single dose of 1.0 mg/kg as IV infusion over approximately 1 hour q3w for the first 12 Weeks as a part of induction phase followed by maintenance dose of 0.3 mg/kg drug every three weeks until significant clinical progression, occurrence of unacceptable toxicity, or withdrawal of consent. The first administration of MSB0010445 was performed 3 days after the last dose of SBRT to the targeted reference lesion. SBRT was administered using a dose and schedule recommended based upon the data showing the best abscopal effect using multiple fractions. If one site was targeted subject received 3 fractions (1 per day) of 8 Gy each (total: 24 Gy). If the target lesion was located in the thorax, the maximum total dose administered was 18 Gy (3 x 6 Gy).
- MSB0010445 High Dose Cohort 1.8 mg/kg: MSB0010445 was administered at a single dose of 1.8 mg/kg as IV infusion over approximately 1 hour q3w for the first 12 Weeks as a part of induction phase followed by maintenance dose of 0.3 mg/kg drug every three weeks until significant clinical progression, occurrence of unacceptable toxicity, or withdrawal of consent. The first administration of MSB0010445 was performed 3 days after the last dose of SBRT to the targeted reference lesion. SBRT was administered using a dose and schedule recommended based upon the data showing the best abscopal effect using multiple fractions. If one site was targeted subject received 3 fractions (1 per day) of 8 Gy each (total: 24 Gy). If the target lesion was located in the thorax, the maximum total dose administered was 18 Gy (3 x 6 Gy).
- MSB0010445 High Dose Cohort 2.4 mg/kg: MSB0010445 was administered at a single dose of 2.4 mg/kg as IV infusion over approximately 1 hour q3w for the first 12 Weeks as a part of induction phase followed by maintenance dose of 0.3 mg/kg drug every three weeks until significant clinical progression, occurrence of unacceptable toxicity, or withdrawal of consent. The first administration of MSB0010445 was performed 3 days after the last dose of SBRT to the targeted reference lesion. SBRT was administered using a dose and schedule recommended based upon the data showing the best abscopal effect using multiple fractions. If one site was targeted subject received 3 fractions (1 per day) of 8 Gy each (total: 24 Gy). If the target lesion was located in the thorax, the maximum total dose administered was 18 Gy (3 x 6 Gy).
Period: Overall Study
Arm/Group | MSB0010445 Low Dose Cohort 0.3 mg/kg | MSB0010445 Intermediate Dose Cohort 1.0 mg/kg | MSB0010445 High Dose Cohort 1.8 mg/kg | MSB0010445 High Dose Cohort 2.4 mg/kg
Started | 2 | 2 | 6 | 2
Completed | 2 | 2 | 6 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analyst set included all subjects who signed informed consent, were enrolled into the study and received at least 1 dose of MSB0010445.
Groups:
- MSB0010445 Low Dose Cohort 0.3 mg/kg: MSB0010445 was administered at a dose of 0.3 mg/kg as IV infusion over approximately 1 hour q3w until significant clinical progression, occurrence of unacceptable toxicity, or withdrawal of consent. The first administration of MSB0010445 was performed 3 days after the last dose of SBRT to the targeted reference lesion. SBRT was administered using a dose and schedule recommended based upon the data showing the best abscopal effect using multiple fractions. One site was targeted and was received 3 fractions (1 per day) of 8 Gy each (total: 24 Gy). If the target lesion was located in the thorax, the maximum total dose was 18 Gy (3 x 6 Gy).
- MSB0010445 Intermediate Dose Cohort 1.0 mg/kg: MSB0010445 was administered at a dose of 1.0 mg/kg as IV infusion over approximately 1 hour q3w until significant clinical progression, occurrence of unacceptable toxicity, or withdrawal of consent. The first administration of MSB0010445 was performed 3 days after the last dose of SBRT to the targeted reference lesion. SBRT was administered using a dose and schedule recommended based upon the data showing the best abscopal effect using multiple fractions. One site was targeted and was received 3 fractions (1 per day) of 8 Gy each (total: 24 Gy). If the target lesion was located in the thorax, the maximum total dose was 18 Gy (3 x 6 Gy).
- MSB0010445 High Dose Cohort 1.8 mg/kg: MSB0010445 was administered at a dose of 1.8 mg/kg as IV infusion over approximately 1 hour q3w until significant clinical progression, occurrence of unacceptable toxicity, or withdrawal of consent. The first administration of MSB0010445 was performed 3 days after the last dose of SBRT to the targeted reference lesion. SBRT was administered using a dose and schedule recommended based upon the data showing the best abscopal effect using multiple fractions. One site was targeted and was received 3 fractions (1 per day) of 8 Gy each (total: 24 Gy). If the target lesion was located in the thorax, the maximum total dose was 18 Gy (3 x 6 Gy).
- MSB0010445 High Dose Cohort 2.4 mg/kg: MSB0010445 was administered at a dose of 2.4 mg/kg as IV infusion over approximately 1 hour q3w until significant clinical progression, occurrence of unacceptable toxicity, or withdrawal of consent. The first administration of MSB0010445 was performed 3 days after the last dose of SBRT to the targeted reference lesion. SBRT was administered using a dose and schedule recommended based upon the data showing the best abscopal effect using multiple fractions. One site was targeted and was received 3 fractions (1 per day) of 8 Gy each (total: 24 Gy). If the target lesion was located in the thorax, the maximum total dose was 18 Gy (3 x 6 Gy).
- Total: Total of all reporting groups
Arm/Group | MSB0010445 Low Dose Cohort 0.3 mg/kg | MSB0010445 Intermediate Dose Cohort 1.0 mg/kg | MSB0010445 High Dose Cohort 1.8 mg/kg | MSB0010445 High Dose Cohort 2.4 mg/kg | Total
Number analyzed (Participants) | 2 | 2 | 6 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.12 (13.48) | 59.55 (4.11) | 59.67 (6.29) | 53.78 (20.03) | 57.91 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 1 | 5
  Male | 1 | 1 | 4 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least 1 Dose Limiting Toxicity (DLT)
Description: DLT was defined as any Grade>= 3 toxicity related to drug, occurring during 21 days post first dose of drug except Grade 3 infusion-related adverse reaction resolving within 6 hours and Transient (<=6 hours) Grade 3 flu-like symptoms/fever controlled with medical management; Transient (<= 24 hours) Grade 3 fatigue, local reactions, headache, nausea, emesis that resolved to <= Grade 1; Grade 3 skin toxicity ,Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 8 x upper limit of normal (ULN)/total bilirubin < 5 x ULN resolving to <= Grade 1 in <7 days after medical management; Grade 3 diarrhea controlled with maximal medical management within 72 hours; Grade 4 lymphopenia that resolves to <= Grade 1 within 7 days & with no clinical manifestations; Grade 3 lab abnormality with no clinical correlation and resolves to <= Grade 1 within 7 days with adequate medical management Tumor flare defined as local pain, irritation or rash localized at sites of known/suspected tumor.
Time Frame: Baseline up to Day 21
Population: Safety analysis set included all subjects who signed informed consent, were enrolled into the study and received at least 1 dose of MSB0010445.
Measure: Number; unit: subjects
Groups:
- MSB0010445 Low Dose Cohort 0.3 mg/kg: MSB0010445 was administered at a single dose of 0.3 mg/kg as IV infusion over approximately 1 hour q3w for the first 12 Weeks as a part of induction phase followed by maintenance dose of 0.3 mg/kg drug every three weeks until significant clinical progression, occurrence of unacceptable toxicity, or withdrawal of consent. The first administration of MSB0010445 was performed 3 days after the last dose of SBRT to the targeted reference lesion. SBRT was administered using a dose and schedule recommended based upon the data showing the best abscopal effect using multiple fractions. If one site was targeted subject received 3 fractions (1 per day) of 8 Gy each (total: 24 Gy). If the target lesion was located in the thorax, the maximum total dose administered was 18 Gy (3 x 6 Gy).
Arm/Group | MSB0010445 Low Dose Cohort 0.3 mg/kg | MSB0010445 Intermediate Dose Cohort 1.0 mg/kg | MSB0010445 High Dose Cohort 1.8 mg/kg | MSB0010445 High Dose Cohort 2.4 mg/kg
Number analyzed (Participants) | 2 | 2 | 6 | 2
subjects | 0 | 0 | 1 | 0

2. Secondary Outcome: Number of Subjects With Best Overall Response (BOR) According to Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1
Description: BOR was defined as a confirmed complete response (CR) or partial response (PR) during second-line treatment. For target lesions (TLs), CR was defined as the disappearance of all TLs, and PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the baseline SLD. For non-target lesions (NTLs), CR was defined as the disappearance of all NTLs and normalization of tumor marker levels.
Time Frame: Screening up to 28 days after last dose of drug; assessed up to maximum of 1.41 years
Population: Safety analysis set included all subjects who signed informed consent, were enrolled into the study and received at least 1 dose of MSB0010445. Here "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Number; unit: subjects
Arm/Group | MSB0010445 Low Dose Cohort 0.3 mg/kg | MSB0010445 Intermediate Dose Cohort 1.0 mg/kg | MSB0010445 High Dose Cohort 1.8 mg/kg | MSB0010445 High Dose Cohort 2.4 mg/kg
Number analyzed (Participants) | 2 | 1 | 4 | 1
subjects
  CR | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (AEs) or Serious AEs
Description: TEAE was defined as an AE that started on or after the first administration of SBRT. An SAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/ significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Time Frame: Screening up to 28 days after last dose of drug; assessed up to maximum of 1.41 years
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | MSB0010445 Low Dose Cohort 0.3 mg/kg | MSB0010445 Intermediate Dose Cohort 1.0 mg/kg | MSB0010445 High Dose Cohort 1.8 mg/kg | MSB0010445 High Dose Cohort 2.4 mg/kg
Number analyzed (Participants) | 2 | 2 | 6 | 2
subjects
  Treatment Emergent Adverse Events | 2 | 2 | 6 | 2
  Serious AEs | 0 | 0 | 3 | 1

ADVERSE EVENTS:
Time Frame: Signing of the informed consent up to 1.41 years
Arm/Group | MSB0010445 Low Dose Cohort 0.3 mg/kg | MSB0010445 Intermediate Dose Cohort 1.0 mg/kg | MSB0010445 High Dose Cohort 1.8 mg/kg | MSB0010445 High Dose Cohort 2.4 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 3/6 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSB0010445 Low Dose Cohort 0.3 mg/kg (N=2) | MSB0010445 Intermediate Dose Cohort 1.0 mg/kg (N=2) | MSB0010445 High Dose Cohort 1.8 mg/kg (N=6) | MSB0010445 High Dose Cohort 2.4 mg/kg (N=2)
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSB0010445 Low Dose Cohort 0.3 mg/kg (N=2) | MSB0010445 Intermediate Dose Cohort 1.0 mg/kg (N=2) | MSB0010445 High Dose Cohort 1.8 mg/kg (N=6) | MSB0010445 High Dose Cohort 2.4 mg/kg (N=2)
Pyrexia (General disorders) | 1 | 0 | 3 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 4 | 0
Influenza like illness (General disorders) | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Depressive symptom (Psychiatric disorders) | 0 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Conjunctival Irritation (Eye disorders) | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Radiation associated pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Early satiety (General disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to sponsor's decision to discontinue the development of MSB0010445. The decision to discontinue development of MSB0010445 was not related to any safety or efficacy concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No